CLINICAL TRIAL: NCT06992869
Title: Matching Mental Health Support to the Needs of People Affected by Parkinson's: Patient and Cost Benefits
Brief Title: Mental Health Support for People Affected by Parkinson's
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: UEA Health Economics Consulting (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 157987; H-2202 (Other Grant/Funding Number: Parkinson's UK)
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease (PD)

STUDY DESIGN:
Intervention Model Description: The intervention uses a wait-list control condition. All participants are on a wait list for 8 weeks before the start of the intervention, which lasts for 8 weeks, and are then followed up 8 weeks afterwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-based psychological therapy (Experimental)
  Interventions: Behavioral: Group-based psychological therapy

INTERVENTIONS:
Behavioral: Group-based psychological therapy — Group-based psychological therapy for (1) adjusting to diagnosis; (2) Parkinson's anxiety and/or depression; and (3) Parkinson's-related cognitive decline

SUMMARY:
In addition to increasingly severe physical symptoms, Parkinson's can cause distressing mental health issues. These include anxiety, depression, and memory and thinking problems, caused by a combination of biological and psychological factors. They can be more disabling than physical symptoms, reduce quality of life and increase risk of mortality. They are also upsetting for family members and unpaid carers, and may necessitate transfer to institutional care. They also increase NHS costs because of expensive hospital admissions. Despite this, there are few specialist mental health professionals or psychological interventions available to help people with Parkinson's.

This study will address this by developing an effective programme of evidence-based psychological interventions for mental health issues in Parkinson's that can be easily delivered by non-experts. Parkinson's mental health specialists at UCL Queen Square Institute of Neurology will work with people affected by Parkinson's and non-psychology health professionals to design specialist interventions for three key mental health needs in Parkinson's, targeted at distinct stages:

1. Adjusting to diagnosis; empowering people to feel more in control.
2. Anxiety and/or depression; using cognitive-behavioural therapy techniques to improve mood, with particular focus on Parkinson's-specific concerns.
3. Advanced Parkinson's; helping people with Parkinson's and those around them to improve management of memory and thinking problems.

The research team will design companion booklets for participants, summarizing each session. The treatment will be piloted for one year. If the interventions prove beneficial to participants and are cost-effective, the resources will be made immediately available to healthcare staff across the UK to improve access to specialist psychological services.

ELIGIBILITY:
All participants will be recruited from the National Hospital for Neurology and Neurosurgery, Queen Square, London.

Inclusion Criteria:

1. Diagnosis of Parkinson's AND

   1. within three years of diagnosis OR
   2. anxiety/depression, as judged by scores above clinical cut-offs on standardized measures OR
   3. developing Parkinson's-related cognitive impairment/hallucinations/delusions, but retaining capacity to consent, as judged by their medical consultant.
2. Aged 18 years and above
3. Sufficiently fluent in English
4. Able to give informed consent
5. Able to attend Queen Square for the intervention
6. Able to complete the self-report questionnaires

Exclusion Criterion:

* Already participating in psychological therapy or research aimed at improving psychological wellbeing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
GAD-7 | Change in GAD-7 scores after 8 weeks of intervention
  Standardized measure of anxiety
PHQ-9 | Change in PHQ-9 scores after 8 weeks of intervention
  Standardized measure of depression
PDQ-39 | Change in PDQ-39 scores after 8 weeks of intervention
  Standardized measure of quality of life in Parkinson's disease
Brief-COPE | Change in Brief-COPE scores after 8 weeks of intervention
  Standardized measure of coping

SECONDARY OUTCOMES:
Healthcare resource use | Change in CSRI healthcare use after 8 weeks of intervention
  Use of healthcare resources as measured by Client Service Receipt Inventory (CSRI)
Acceptability | Following the 8 week intervention
  Quantitative indicator of acceptability, as measured by Likert scales on questionnaire
Acceptability | Following the 8 weeks of intervention
  Qualitative indicator of acceptability from thematic analysis of open-ended questions on questionnaires and focus group interviews
Ease of delivery by non-experts | Following 8-weeks of intervention
  Ease of delivery by non-experts, determined by comparing change in GAD-7 by intervention lead (nurse vs psychologist)
Ease of delivery by non-experts | Following 8-weeks of intervention
  Ease of delivery by non-experts, determined by comparing change in PHQ-9 by intervention lead (nurse vs psychologist)
Ease of delivery by non-expert | Following 8-weeks of intervention
  Ease of delivery by non-expert, as determined by comparing chnage in PDQ-39 by intervention lead (nurse vs psychologist)
Ease of delivery by non-expert | Following 8-weeks of intervention
  Ease of delivery by non-expert, as determined by comparing change in Brief-COPE by intervention lead (nurse vs psychologist)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Foley, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not have explicit consent for sharing of IPD at present.